CLINICAL TRIAL: NCT00138645
Title: The Effects of Formula Diet on Body Weight, Body Composition, and Biomarkers for Disease Compared to a Standard Diet
Acronym: FORMULA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Sunny Health Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Corby K. Martin, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 25004
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MicroDiet (Experimental): Participants randomized to the MicroDiet group (1200 kcal/day) will be instructed by a Registered Dietitian to consume (one shake and 3 cookies; 240 kcal) for two meals each day for Months 1 through 3. They will be provided with meal plans for the meal that they do not replace with MicroDiet. During Months 4 through 6, participants in the MicroDiet group will be instructed to replace one meal per day with MD (the energy content of the meal plan will still be 1200 kcal/day). Participants will also be encouraged to eat or drink MD for snacks. The rest of the diet will consist of healthy foods, as outlined above. To help participants adhere to the MicroDiet regimen, they will meet with a registered dietitian for one hour at Week 0 and 30 minutes at Weeks 2 and 4, and every month thereafter.
  Interventions: Behavioral: MicroDiet
- Healthy Diet (Active Comparator): Participants randomized to the Healthy Diet group will be prescribed a traditional food-based diet that contains the same number of kilocalories (1200/day) as the MicroDiet. The Healthy Diet will consist of the same foods that are used in the meal plans for the MicroDiet group. The Healthy Diet group will be instructed not to use meal replacements such as shakes (e.g., Slim Fast®), nutrition bars (e.g., Balance Bar®), or portion-controlled meals (e.g., Healthy Choice entrees).
  Interventions: Behavioral: Healthy Diet

INTERVENTIONS:
Behavioral: MicroDiet — MicroDiet
  Arms: MicroDiet
Behavioral: Healthy Diet — Participants randomized to the Healthy Diet group will be prescribed a traditional food-based diet that contains the same number of kilocalories (1200/day) as the MicroDiet but will be instructed not to use meal replacements
  Arms: Healthy Diet

SUMMARY:
It is hypothesized that the use of a partial supplement diet, which includes the use of meal replacements, will result in significantly greater weight loss after three and six months compared to an isocaloric diet that does not include supplements. It is also hypothesized that the partial supplement diet will result in larger improvements in body composition, disease biomarkers, and health parameters (blood pressure, lipids) compared to the non-supplement diet. Finally, it is hypothesized that subjective ratings of satiety will be significantly higher, and ratings of hunger lower, in the group consuming a partial supplement diet.

DETAILED DESCRIPTION:
In recent decades, the prevalence of overweight and obesity has increased dramatically in developed countries. Obesity is associated with diseases such as diabetes, cardiovascular disease, hypertension, and certain cancers. Modest amounts of weight loss (e.g., 5% to 10% of initial body weight) significantly improve health and improve disease status. Recent evidence suggests that the use of supplements or meal replacements promotes greater weight loss than isocaloric food-based diets. In addition, diets that are high in protein are associated with greater ratings of satiety and reduced food intake, as well as greater weight loss, compared to lower protein diets.

The purpose of the proposed study is to test the effect of a partial supplement diet on body weight, body composition, and biomarkers for disease compared to an isocaloric diet that consists of a traditional food-based meal plan. Overweight and obese (BMI 25 to 35) participants will participate in this six-month study. The primary outcome variable is body weight loss and the secondary outcome variables include body composition, blood pressure, lipids, and subjective ratings of satiety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender; of all ethnic backgrounds.
* Healthy person who has not been diagnosed with diabetes, cardiovascular illness, renal, hepatic or other chronic diseases
* > 17 years and < 66 years of age
* Body mass index (BMI; kg/m2) between 25 and 35
* For females with the potential to bear children, they meet one of the following criteria:

  * They are willing to use an acceptable method of birth control (e.g., oral contraceptive tablets, implanted contraceptive hormones, Depo-Provera® contraceptive injections, intrauterine devices, prophylactic condoms with spermicide, contraceptive diaphragms with spermicide, cervical caps with spermicide), or are in a monogamous relationship with a partner who has had a vasectomy.
  * They are sexually abstinent and intend to continue this practice, at least for the duration of the study.

Exclusion Criteria:

* > 65 years and < 18 years of age
* Regular use of medications other than birth control, vitamins or hormone replacement therapy
* Diabetes mellitus (fasting blood sugar [FBS] > 126); persons with impaired glucose tolerance (FBS 100-125) may be admitted to the study.
* Use of tobacco products
* Depression or mental illness requiring treatment or medication within the last six months
* For women, pregnancy, breast feeding, postpartum < 6 months, planning a pregnancy during the study, or are not using an acceptable method of contraception
* Use of medications or herbal supplements that affect appetite or body weight for the previous three months
* Patients requiring restriction of protein intake
* Impaired kidney function (creatinine > 1.5) or liver function (liver enzymes > 3 times the upper limits of normal)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K. Martin, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Diet: Healthy Diet
Period: Overall Study
Arm/Group | MicroDiet | Healthy Diet
Started | 30 | 30
Completed | 24 | 23
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MicroDiet | Healthy Diet | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11.4) | 43 (11.4) | 42 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Body Weight Loss (kg and Percent) at Months 3 and 6
Time Frame: April 2005 to May 2006
Reporting Status: Not Posted

2. Secondary Outcome: Change in Body Composition at Months 3 and 6
Time Frame: April 2005 to May 2006
Reporting Status: Not Posted

3. Secondary Outcome: Disease Biomarkers (Cholesterol, Triglycerides, Etc.) at Months 3 and 6
Time Frame: April 2005 to May 2006
Reporting Status: Not Posted

4. Secondary Outcome: Subjective Ratings of Appetite at Week 2 and Months 1, 2, 3, 4, 5, and 6
Time Frame: April 2005 to May 2006
Reporting Status: Not Posted

5. Primary Outcome: Percent Change in Body Weight (Completers).
Description: Percent change in body weight from baseline to week 24(completers).
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: change in percent:baseline body weight
Arm/Group | MicroDiet | Healthy Diet
Number analyzed (Participants) | 24 | 23
change in percent:baseline body weight | 7.3 (1.3) | 7.0 (1.3)

ADVERSE EVENTS:
Groups:
- MicroDiet: Participants randomized to the MicroDiet
- Healthy Diet: participants randomized to the low-calorie diet.
Arm/Group | MicroDiet | Healthy Diet
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No